CLINICAL TRIAL: NCT05203029
Title: Effectiveness of Aerobic Exercises and Laughter Yoga Compared With Yoga in Anxiety and Depression Levels of Breast Cancer Survivors; a Double-blind Three Arm Clinical Trial Study
Brief Title: Effectiveness of Aerobic Exercises and Laughter Yoga Compared With Yoga in Anxiety/Depression Levels in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fateme Abedini, Principal investigator, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 55516
Record Dates: First submitted 2022-01-12; First posted 2022-01-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer Survivors
Keywords: Aerobic exercises; Laughter yoga; Yoga; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercises (Experimental): The warm-up for 5 minutes; stretching exercises include stretching the neck to the sides, stretching the muscles of the shoulder girdle, back, and legs for 10 minutes; resistance exercises for 15 minutes, which will initially be applied in a light and weight-bearing manner, and in each session, according to the patient's progress, using free lightweights; light aerobic exercise for 10 minutes standing, sitting and lying down by controlling patients' heartbeat; cool down for 5 minutes.
  Interventions: Other: Online exercise
- Laughter yoga (Experimental): Breathing techniques for 20 minutes including deep breathing, diaphragmatic breathing, tap on immune-boosting centers like thymus; laughter concert for 20 minutes such as laughter for no reason, childish movements, release the inner child; and laughter meditation for 5 minutes.
  Interventions: Other: Online exercise
- Yoga (Active Comparator): Meditation and deep breathing for 10 minutes; physical posture for 15 minutes; 15 minutes relaxation exercises; and 5 minutes mindfulness practices.
  Interventions: Other: Online exercise

INTERVENTIONS:
Other: Online exercise — Patients in each group will be added to the specific group on Whatsapp, and the schedule and information about the exercise will be explained there. Furthermore, patients will be joined to particular pages on Instagram, and exercises will be performed through Live on that pages. All the patients will exercise for 12 weeks, two or three times every week.

SUMMARY:
90% of breast cancer survivors experience cancer-related fatigue which decreases the physical activity. Moreover, due to the cancer treatments depression and anxiety will be happened. Previous studies showed the effect of physical activity on reduction of depression and anxiety; therefore the aim of this study is to evaluate the effectiveness of aerobic exercises and laughter yoga compared with yoga in anxiety and depression levels in breast cancer survivors.

DETAILED DESCRIPTION:
204 breast cancer survivors will be randomized to each of these three groups: Group 1, 12 weeks aerobic exercises; Group 2, 12 weeks of laughter yoga; and Group 3, 12 weeks of yoga.

To assess the effectiveness of these exercises in depression and anxiety levels, patients will complete the hospital anxiety and depression scale (HADS) questionnaire before and after the 3-month exercise.

For secondary outcomes, patients will complete the following questionnaires before and after the 3-month exercise: 36-item short-form survey (SF-36), Minnesota Living with Heart Failure Questionnaire (MLHFQ), Insomnia Severity Index, Beck's depression inventory-Ⅱ (BDI-Ⅱ), Chalder's chronic fatigue syndrome, and five facet mindfulness questionnaire (FFMQ).

The effectiveness of the mentioned exercises in primary and secondary outcomes will be assessed using ANOVA/ANCOVA analysis by adjusting the baseline assessment. Mean difference (MD) and standardized mean difference (SMD) with their 95% confidence interval (CI) will be reported to show the effectiveness of aerobic exercises and laughter yoga compared with yoga in different outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 to 65 years
* Patients with stage Ⅰ-Ⅲ of breast cancer
* Chemotherapy is completed at least six months before registration
* Lack of active participation in regular exercise programs

Exclusion Criteria:

* Reluctance to cooperate and enter the study
* Do not complete the questionnaires correctly
* Have diseases such as severe heart failure (Minnesota Living with Heart Failure Questionnaire score more than 50), severe valvular disease, coronary stenosis of the heart, and metastatic cancer
* Feel chest pain and dizziness during the exercise
* Patients currently receiving treatment
* Patients who do not have the physical ability to participate in the exercise
* Patients with mental health disorders that cannot participate in the exercise

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Changes in the anxiety and depression levels after twelve weeks of exercises | 0 and 3 months
  Hospital anxiety and depression scale (HADS) questionnaire will be used to determine the anxiety and depression levels. This questionnaire contains 14 questions, of which seven concern anxiety and seven concern depression. Each question is scored from 0 (never) to 3 (almost always); the final score will be 0 to 52, and the higher scores indicate greater anxiety and depression.

SECONDARY OUTCOMES:
Changes in the general quality of life after twelve weeks of exercises | 0 and 3 months
  36-item short form survey (SF-36) questionnaire will be used to determine the quality of life. This questionnaire comprises 36 items and eight domains, including limitations in physical activities because of health problems, limitations in social activities because of physical or emotional issues, limitations in usual role activities because of physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities because of emotional problems, vitality (energy and fatigue), and general health perceptions. Each question is scored from 0 to 100; the final score is the average score from 0 to 100, and the higher scores show a better quality of life. The scores will be reported for each domain separately
Changes in the disease-specific quality of life after twelve weeks of exercises | 0 and 3 months
  Minnesota Living with Heart Failure Questionnaire (MLHFQ) will be used to determine the disease-specific quality of life. It has 21 items in physical, emotional and socioeconomic dimensions; each item scored from 0 to 5 provides a total score between 0 to 105: the higher the score, the lower quality of life.
Changes in the Insomnia severity after twelve weeks of exercises | 0 and 3 months
  The Insomnia Severity Index questionnaire will be used to determine the insomnia severity. It has seven questions; each item has a score from 0 to 4. The seven answers are added up to get a total score from 0 to 28. The higher scores represent severe insomnia.
Changes in depression after twelve weeks of exercises | 0 and 3 months
  Beck's depression inventory-Ⅱ (BDI-Ⅱ) will be used to measure depression. This questionnaire has 21 questions scored from 0 to 3. The total score will calculate by adding up all the scores-the higher scores indicating the higher depression.
Changes in chronic fatigue after twelve weeks of exercises | 0 and 3 months
  Chalder's chronic fatigue syndrome questionnaire will be utilized to measure chronic fatigue. This questionnaire has 14 items, eight items are about physical symptoms, and six other items are about mental symptoms. Each question scored between 0 to 3, and the total score will be 0 to 42. The higher the score, the more suffer from fatigue.
Changes in mindfulness after twelve weeks of exercises | 0 and 3 months
  Mindfulness will be measured by five facet mindfulness questionnaire (FFMQ). It has 39 questions in five domains: observation, description, aware actions, non-judgmental inner experience, and non-reactivity. Each question scored between 1 to 5, and the total score will be in the range of 39 to 195. The higher score shows the higher mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Fateme Abedini, MSc, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Isfahan University of Medical Sciences, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No